CLINICAL TRIAL: NCT01614938
Title: Phase II Trial of Docetaxel-Cisplatin Neoadjuvant Chemotherapy Followed by Concurrent Radiotherapy With Cetuximab or Weekly Cisplatin in Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Induction Chemotherapy Followed by Concurrent Radiation With Cetuximab or Cisplatin in Locally Advanced Nasopharyngeal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guo-Pei Zhu, M.D., Associated Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HN201002
Record Dates: First submitted 2012-06-05; First posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Locally advanced; Cetuximab; Weekly cisplatin chemotherapy; Intensity-modulated radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cetuximab; Cisplatin; Docetaxel; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cisplatin-radiotherapy (CRT) (Active Comparator): The arm receiving docetaxel-cisplatin neoadjuvant chemotherapy followed by concurrent weekly cisplatin and radiotherapy
  Interventions: Drug: Docetaxel; Radiation: Intensity-modulated radiotherapy; Drug: Cisplatin
- cetuximab-radiotherapy (ERT) (Experimental): The arm receiving docetaxel-cisplatin neoadjuvant chemotherapy followed by concurrent cetuximab and radiotherapy
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: Docetaxel; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Cetuximab — 400 mg/m2 initial dose before radiation, then 250 mg/m2 weekly during radiation
  Other Names: Erbitux
  Arms: cetuximab-radiotherapy (ERT)
Drug: Cisplatin — 2 cycles of induction chemotherapy every 3 weeks with cisplatin 80 mg/m2 D1-3
  Other Names: Platinol
  Arms: cetuximab-radiotherapy (ERT)
Drug: Docetaxel — 2 cycles of induction chemotherapy every 3 weeks with docetaxel 75 mg/m2 D1
  Other Names: Taxotere
Radiation: Intensity-modulated radiotherapy — a total dose of 66-70.4Gy in 30-32 fractions over 6-6.5 weeks planned to be delivered to the PTV of gross tumor
  Other Names: IMRT
Drug: Cisplatin — 2 cycles of induction chemotherapy every 3 weeks with cisplatin 80 mg/m2 D1-3, then 6 cycles of concomitant chemotherapy every week with cisplatin 30 mg/m2 D1
  Other Names: Platinol
  Arms: cisplatin-radiotherapy (CRT)

SUMMARY:
The purpose of this study is to compare the efficacy and toxicity of docetaxel-cisplatin neoadjuvant chemotherapy followed by concurrent radiotherapy with cetuximab or weekly cisplatin in locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Although concurrent chemoradiation is the standard treatment modality for locally advanced nasopharyngeal carcinoma (NPC), high incidences of distant metastases and severe treatment related toxicities have become an obstacle to be overcome. A phase Ⅱ study conducted by Hui et al. showed that neoadjuvant docetaxel-cisplatin (TP) chemotherapy followed by concurrent chemoradiotherapy was superior to the standard concomitant chemoradiation in terms of the 3-year OS without significantly exacerbating the acute toxicities. Moreover, Bonner et al. demonstrated that RT with concurrent Cetuximab significantly improved the 5-year OS and did not increase the treatment induced toxicities when compared with RT alone. Therefore, we initiated this study to compare the efficacy and toxicity of the two regimens, neoadjuvant chemotherapy followed by concurrent radiotherapy with cetuximab or weekly cisplatin for locally advanced NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven nasopharyngeal carcinoma (WHO type 2 or 3)
2. Stage Ⅲ-ⅣB disease (AJCC/UICC 2009)
3. ECOG performance status of 0-1
4. Life expectancy of more than 6 months
5. Signed written informed consent
6. Adequate organ function including the following:

   * Absolute neutrophil count (ANC) >= 1.5 * 109/l
   * Platelets count >= 100 * 109/l
   * Hemoglobin >= 10 g/dl
   * AST and ALT <= 2.5 times institutional upper limit of normal (ULN)
   * Total bilirubin <= 1.5 times institutional ULN
   * Creatinine clearance >= 50 ml/min
   * Serum creatine <= 1 times ULN

Exclusion Criteria:

1. Evidence of distant metastasis
2. Prior chemotherapy or anti-cancer biologic therapy for any type of cancer, or prior radiotherapy to the head and neck region
3. Other previous or concomitant cancer, except for in situ cervical cancer and cutaneous basal cell carcinoma
4. Pregnant or breast-feeding females, or females and males of childbearing potential not taking adequate contraceptive measures
5. Presence of an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 3 years
  The time from date of randomization until date of first documented disease progression or death from any cause, assessed up to 3 years.

SECONDARY OUTCOMES:
Overall survival | up to 3 years
  The time from date of randomization until date of death due to any cause, assessed up to 3 years.
Locoregional recurrence-free survival | up to 3 years
  The time from date of randomization until date of first documented disease recurrence at a locoregional site, assessed up to 3 years.
Distant metastasis-free survival | up to 3 years
  The time from date of randomization until date of first documented distant metastasis, assessed up to 3 years.
Number of participants with hematologic toxicity events occurred during two cycles of neoadjuvant chemotherapy according to CTCAE v4.0 | 1, 2, 3 weeks post-dose
Number of participants with acute toxicities (hematologic toxicity events, oral mucositis, acne-like rash) occurred during the concurrent treatment according to CTCAE v4.0 | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
Number of participants with late toxicities (hematologic toxicity events, dysphagia, acne-like rash) occurred from 3 months after completion of radiotherapy to last follow-up visit according to CTCAE v4.0 | Every 3 months during the first 2 years, then every 6 months during year 3 after completion of radiotherapy
Score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Core 35 (EORTC QLQ-HN35) during the concurrent treatment | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  QoL score will be documented on each weekend during the course of radiotherapy
Score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Core 35 (EORTC QLQ-HN35) at 3 months after completion of radiotherapy | At 3 months after completion of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Zhu, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xu T, Liu Y, Dou S, Li F, Guan X, Zhu G. Weekly cetuximab concurrent with IMRT aggravated radiation-induced oral mucositis in locally advanced nasopharyngeal carcinoma: Results of a randomized phase II study. Oral Oncol. 2015 Sep;51(9):875-9. doi: 10.1016/j.oraloncology.2015.06.008. Epub 2015 Jul 7. PMID 26163437